CLINICAL TRIAL: NCT04443426
Title: Modulation of Circulating Levels of the Ketone Body 3-hydroxybutyrate in Patients With Chronic Heart Failure: Cardiovascular Effects
Acronym: KETO-KINETICS1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KETO- CHF 1-10-72-362-18
Record Dates: First submitted 2019-05-20; First posted 2020-06-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure; Ketosis; Ketonemia
Keywords: Metabolism
MeSH Terms: conditions — Heart Failure; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose oral 3-hydroxybutyrate monoester (Experimental): Cross-over study in 8 patients receiving single-dose oral 3-hydroxybutyrate monoester, 3-OHB salt and placebo.
  Interventions: Dietary Supplement: Ketone Monoester
- Single dose oral 3-hydroxybutyrate Salt (Experimental)
  Interventions: Dietary Supplement: Oral 3-hydroxybutyrate salts
- Single dose oral placebo (Placebo Comparator): maltodextrin-based, isocaloric to ketone dosis.
  Interventions: Dietary Supplement: Carbohydrate Placebo

INTERVENTIONS:
Dietary Supplement: Oral 3-hydroxybutyrate salts — Comercially available 3-hydroxybutyrate salts with 36 grams of 3-OHB salts three times daily.
  Arms: Single dose oral 3-hydroxybutyrate Salt
Dietary Supplement: Carbohydrate Placebo — Comercially available carbohydrate sports drink. The placebo dose is isocaloric to the 3-hydroxy butyrate dose.
  Arms: Single dose oral placebo
Dietary Supplement: Ketone Monoester — Commercially available ketone monoester in a dosage isocaloric to 3-OHB salts.
  Arms: Single dose oral 3-hydroxybutyrate monoester

SUMMARY:
The ketone body 3-hydroxybutyrate (3-OHB) is a naturally occurring energy substrate, and is associated with increased life span and improved health. We have previously shown that intravenous 3-OHB treatment increases myocardial blood flow > 70% in healthy humans and data from our group show that 3-OHB increases cardiac output by 40 % in patients with heart failure.

In this study the investigators aim to investigate:

1. If this effect is reproducible with a commercially available oral ketone supplements
2. The safety of commercially available ketone supplements in heart failure patients

DETAILED DESCRIPTION:
Heart Failure (HF) is a major public health issue because the disease affects 1-2% of the Western population and the lifetime risk of HF is 20%. HF is responsible for 1-2% of all healthcare expenditures. Despite major improvements in the management and care of patients with HF, the 1-year mortality in patients with HF is 13 % and >50% of HF-patients is admitted during a 2.5 year period. Furthermore patients with HF have markedly decreased physical capacity and quality of life. Thus, there is a need for new treatment modalities in this group of patients.

Ketone bodies are produced in the liver and are of vital importance in the human body for energy generation in the heart and brain during fasting, exercise and severe illness. Ketosis can be safely obtained using dietary supplements and can increase exercise capacity in athletes. The most important ketone bodies are 3-hydroxybutyrate (3-OHB) and acetoacetate. Recently, it was demonstrated that patients with severe HF have increased myocardial utilization of the ketone body 3-hydroxybutyrate.

We have shown, using positron emission tomography, that ketone body infusion reduces myocardial glucose uptake and increases myocardial blood flow in healthy subjects. Data from another study conducted by our group show a 40% increase in cardiac output during infusion of 3-OHB.

Presently there are no data on the clinical cardiovascular and metabolic effects of long-term oral ketone-supplementation in patients with chronic HF.

In this study the investigators will whether ketosis obtained by oral ketone supplements affects hemodynamics and contractile function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure;
* NYHA class II-III
* Left Ventricular Ejection Fraction <40%

Exclusion Criteria:

* Diabetes or HbA1c > 48 mmol/mol
* Significant cardiac valve disease,
* Severe stable angina pectoris
* Severe comorbidity as judged by investigator,
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (L/min) | 5 hours - Area under the curve
  Right Heart Catherization

SECONDARY OUTCOMES:
Left Ventricle Ejection Fraction (%) | 5 Hours - Area under the curve
  Echocardiography
Left Ventricular filling pressure (mmHg) | 5 hours - Area under the curve
  Right Heart Catherization

CONTACTS AND LOCATIONS:
Overall Officials: Kristian H Christensen, MD, Principal Investigator — Aarhus Universitetshospital - Department of Cardiology
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT04443426/Prot_SAP_000.pdf